CLINICAL TRIAL: NCT04029753
Title: Effects of Walking Out From Operating Room on Postoperative Recovery of Patients Undergoing Laparoscopic Radical Gastrectomy
Brief Title: Patients Undergoing Laparoscopic Radical Gastrectomy Walk Out From Operating Room After Surgery ( WOFOR-G-01 )
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, SanQing Jin, professor, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019ZSLYEC-053
Record Dates: First submitted 2019-07-14; First posted 2019-07-23 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Laparoscopic Radical Gastrectomy; Enhanced Recovery After Surgery
Keywords: Early Mobilization

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Walk out from operating room (Experimental): Patients will return to the ward after surgery by walking.
  Interventions: Behavioral: Walk out from operating room
- Leave operating room by transporting bed (No Intervention): Patients will return to the ward after surgery by lying on the transporting bed.

INTERVENTIONS:
Behavioral: Walk out from operating room — After the surgery of laparoscopic radical gastrectomy, patients will be encouraged to walk out from the operating room and return to the ward by walking under the condition of stable physiological parameters, painlessness, clear consciousness and normal muscle strength of lower limb.
  Arms: Walk out from operating room

SUMMARY:
Although early and progressive mobility is widely accepted as an important aspect of postoperative care, guidelines and recommendations suggesting the exact timing and intensity of mobilization efforts are nonexistent. We propose the concept of walking out from the operating room (WOFOR), which means under meticulous anesthesia treatment, perfect postoperative analgesia conditions, rigorous assessment of consciousness and normal muscle strength, postoperative patients can walk safely out of the operating room and return to the ward. The aim of this randomized controlled trial is to investigate the effect of walking out from the operating room on the postoperative recovery of patients undergoing laparoscopic radical gastrectomy.

DETAILED DESCRIPTION:
Postoperative bed rest increases the risk of complications such as thromboembolism and intestinal adhesion, but actual clinical effects of early mobilization still need randomized control trails to prove. The aim of this randomized controlled trial is to investigate the effect of walking out from the operating room (very early mobilization after surgery) on the postoperative recovery of patients undergoing laparoscopic radical gastrectomy.

A sample size of 96 patients in each group is calculated by a prior power analysis on the basis of the following assumptions: (1) an absolute reduction in the length of the hospital stay by 1 day, (2) standard deviations are 2 days in the experimental group and the control group, (3)α=0.05, (4) power 90% and (5) missed follow-up rate 10%. Considering that this study is not for rare diseases, in order to ensure adequate sample size, we adjust the sample size of each group to an integer of 100.

Patients will receive written and verbal information about the trial before written consent is obtained. The randomization will take place when the surgeons confirm preliminarily there is no need to place drainage tube for coelom hyperthermia perfusion after laparoscopy. Then patients will be assigned to either intervention (return to ward by walking) or control group (return to ward by lying on the transporting bed). A stratified randomization with three factors including sex, age and total or distal gastrectomy will be performed to ensure an even spread. The randomization is performed using concealed allocation where envelopes are prepared externally using a randomization list prepared by a statistician.

The patients will receive general anesthesia combined with epidural analgesia. After surgery, the patients will be evaluated whether fulfilling the criteria for mobilization including stable physiological parameters, consciousness, normal level of orientation and muscle strength, and painlessness every ten minutes. If patients fulfill the criteria, they will receive different methods of returning to the ward based on the grouping. In the control group, the patient will return to the ward by lying on the transporting bed. In the intervention group, the patients will be raised to a sitting position for five minutes. If the patients do not complain any discomfort and have stable physiological parameters, they will be encouraged to stand. If standing do not cause any discomfort, they will be encouraged to walk within the range of 5-meter long and 60-centimeter wide. If patients can walk within the range, they will return to the surgical ward by walking under the protection of medical staffs.

Then, all study patients will be subject to the same management such as the guidance of drink and diet recovery, the guidance of mobilization in the ward, nutrition supplement after surgery, and the criteria of drainage removal and hospital discharge. The outcomes such as the length of hospital stay after surgery will be recorded and analyzed to evaluate the effects of walking out from the operating room. The analysis of Intention-to-treat and Per-protocol-sets will be both performed by statisticians.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 Years old
2. scheduled for laparoscopic radical gastrectomy.
3. American Society of Anesthesiologists (ASA) grading I or II

Exclusion Criteria:

1. Patients have severe cardiac diseases (cardiac function grading greater than grade 3/arrhythmia including sick sinus syndrome, atrial fibrillation, atrial flutter, atrioventricular block, frequent ventricular premature,multiple ventricular premature, ventricular premature R on T, ventricular fibrillation and ventricular flutter/acute coronary syndrome) or respiratory failure or hepatic failure or renal failure;
2. Body mass index (BMI) ≥30 kg/m2;
3. Preoperative hemoglobin<80 g/L or albumin<30 g/L
4. Patients have diabetics or patients with gastric emptying disorders;
5. Patients with poor blood pressure control (receive regular antihypertensive medical treatment but still have systolic blood pressure>150 mmHg and/or diastolic blood pressure>90 mmHg );
6. Patients have schizophrenia, epilepsy, Parkinson's disease, mental retardation, or hearing impairment.
7. Patients have thrombosis such as in lower extremity or in vena cava or in other veins.
8. Patients have neuromuscular disorders affecting lower limb activity, such as myasthenia gravis and cerebral infarction, which cause lower limb muscle weakness;
9. Patients have contraindications for epidural puncture.
10. Postoperative placement of drainage tube for coelom hyperthermia perfusion
11. Patients participate in other clinical trials.
12. Patients refuse to sign informed consent for research.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-08-27 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay after surgery | at hospital discharge(expected 7 days after surgery)
  hospital stay time from operation completion to actual hospital discharge

SECONDARY OUTCOMES:
Time to fulfill the criteria of hospital discharge | expected 7 days after surgery
  the ideal time point for discharge, which is also considered as recovery time. The criteria for measuring recovery time included: 1) the patients receive 80% of normal nutritional support （30 kcal/kg/day calories is regard as normal nutritional support）and 30ml/kg fluid intake by oral; 2)gastrointestinal function has been restored: flatus with or without defecation; 3)analgesic-free, which is defined as visual analogue scale ≤3 without intravenous analgesic drugs, 4) adequate mobility without support; 5) afebrile status without major infectious complications
The percentage of patients feeling ready for hospital discharge when they reach the discharge criteria. | expected 6 days after surgery
  the percentage of patients feeling ready for hospital discharge when they reach the discharge criteria.
Postoperative recovery score using 40-item quality of recovery scoring system(QoR-40) | every 24 hours after surgery (at 1-day, 2-day, 3-day), and then every 48 hours until the discharge after surgery (at 5-day, 7-day (if any), 9-day (if any)...)
  to evaluate the postoperative recovery using 40-item quality of recovery scoring system including emotional state (9items), physical comfort (12 items), physical independence (5 items), psychologic support (7 items), and pain (7 items). Each item is graded on a five-point Likert scale, and global scores range from 40 (extremely poor quality of recovery)to 200 (high quality of recovery). Each item is graded on a five-point Likert scale, and global scores range from 40 (extremely poor quality of recovery) to 200 (high quality of recovery).
Six-minute walking test | the day before surgery, every 24 hours after surgery (at 1-day, 2-day, 3-day), and then every 48 hours until the discharge after surgery (at 5-day, 7-day (if any), 9-day (if any)...)
  physical capacity measured with the six-minute Walking test before surgery and after surgery.The longer walking distance in six minutes, the better physical capacity.
Anxiety score | the day before surgery, every 24 hours after surgery (at 1-day, 2-day, 3-day), and then every 48 hours until the discharge after surgery (at 5-day, 7-day (if any), 9-day (if any)...)
  anxiety state evaluated by State-Trait Anxiety Inventory Form. The form used in this study is the Chinese version. The scales consist of 20 items; the responses range from 1 to 4 points (forced choice). The scores range from 20 (extremely low level of anxiety) to 80 (high level of anxiety). The STAI classifies anxiety into five stages: stages 1 and 2 suggest mild anxiety; stage 3 suggests moderate anxiety, and stages 4 and 5 suggest severe anxiety.
Postoperative pain score | every 24 hours after surgery (at 1-day, 2-day, 3-day), and then every 48 hours until the discharge after surgery (at 5-day, 7-day (if any), 9-day (if any)...)
  pain score after surgery is evaluated using a visual analogue scale 0-10 rated by the patients
Severity of postoperative nausea and vomiting | every 24 hours after surgery (at 1-day, 2-day, 3-day)
  everity of postoperative nausea and vomiting is measured with the PONV intensity grading. Briefly, no PONV is defined as the absence of any emetic symptoms and nausea during the entire study period. Mild PONV is defined as the occurrence of mild nausea or one episode of vomiting if caused by an exogenous stimulus such as drinking or movement. Moderate PONV is reached when the patient vomits up to 2 times or experiences nausea that requires a rescue antiemetic therapy only once. Severe PONV is reached if the patient suffers more than two emetic episodes or needs more than one dose of a rescue antiemetic drugs.
Time to first flatus after surgery | from the time of operation completion until the time of the first flatus occurrence, assessed up to 7 days.
  the time length between operation completion and the first flatus
Time to first defecation after surgery | from the time of operation completion until the time of the first defecation occurrence, assessed up to 10 days.
  the time length between operation completion and the first defecation
The volume of drainage after surgery | every 24 hours from the time of operation completion until the time of drainage tube removal, assessed up to 30 days.
  total volume of drainage after surgery and drainage volume every 24 hours after surgery.
Time to the removal of drainage tube | from the time of operation completion until the time of drainage tube removal, assessed up to 30 days.
  recorded the time length between operation completion and the removal of drainage tube
Incidence of surgical complications within 7 days after surgery | 7 days after surgery
  incidence of bleeding, wound infection, wound dehiscence, ileus, stenosis, Leakage within 30 days after surgery
Incidence of surgical complications within 30 days after surgery | 30 days after surgery
  incidence of bleeding, wound infection, wound dehiscence, ileus, stenosis, Leakage within 30 days after surgery
Unplanned re-admission incidence within 30 days after operation | 30 days after operation
  incidence of unplanned admit to hospital again within 30 days after operation
Incidence of major cardiovascular and cerebrovascular adverse events within 30 days after operation | 30 days after operation
  incidence of a complex event consisting of all-cause death, myocardial infarction, stroke and emergency target vessel revascularization within 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sanqing Jin, MD, Principal Investigator — The Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- the Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Ding J, Sun B, Song P, Liu S, Chen H, Feng M, Guan W. The application of enhanced recovery after surgery (ERAS)/fast-track surgery in gastrectomy for gastric cancer: a systematic review and meta-analysis. Oncotarget. 2017 Jun 20;8(43):75699-75711. doi: 10.18632/oncotarget.18581. eCollection 2017 Sep 26. PMID 29088903
- [Background] Mortensen K, Nilsson M, Slim K, Schafer M, Mariette C, Braga M, Carli F, Demartines N, Griffin SM, Lassen K; Enhanced Recovery After Surgery (ERAS(R)) Group. Consensus guidelines for enhanced recovery after gastrectomy: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations. Br J Surg. 2014 Sep;101(10):1209-29. doi: 10.1002/bjs.9582. Epub 2014 Jul 21. PMID 25047143
- [Background] Pedziwiatr M, Mavrikis J, Witowski J, Adamos A, Major P, Nowakowski M, Budzynski A. Current status of enhanced recovery after surgery (ERAS) protocol in gastrointestinal surgery. Med Oncol. 2018 May 9;35(6):95. doi: 10.1007/s12032-018-1153-0. PMID 29744679
- [Background] Mingjie X, Luyao Z, Ze T, YinQuan Z, Quan W. Laparoscopic Radical Gastrectomy for Resectable Advanced Gastric Cancer Within Enhanced Recovery Programs: A Prospective Randomized Controlled Trial. J Laparoendosc Adv Surg Tech A. 2017 Sep;27(9):959-964. doi: 10.1089/lap.2016.0057. Epub 2016 Nov 22. PMID 27875094
- [Background] Chen Hu J, Xin Jiang L, Cai L, Tao Zheng H, Yuan Hu S, Bing Chen H, Chang Wu G, Fei Zhang Y, Chuan Lv Z. Preliminary experience of fast-track surgery combined with laparoscopy-assisted radical distal gastrectomy for gastric cancer. J Gastrointest Surg. 2012 Oct;16(10):1830-9. doi: 10.1007/s11605-012-1969-4. Epub 2012 Aug 2. PMID 22854954
- [Background] Li MZ, Wu WH, Li L, Zhou XF, Zhu HL, Li JF, He YL. Is ERAS effective and safe in laparoscopic gastrectomy for gastric carcinoma? A meta-analysis. World J Surg Oncol. 2018 Jan 26;16(1):17. doi: 10.1186/s12957-018-1309-6. PMID 29373978
- [Background] Ma Z, Bao X, Gu J. Effects of laparoscopic radical gastrectomy and the influence on immune function and inflammatory factors. Exp Ther Med. 2016 Aug;12(2):983-986. doi: 10.3892/etm.2016.3404. Epub 2016 May 27. PMID 27446308
- [Background] Abdikarim I, Cao XY, Li SZ, Zhao YQ, Taupyk Y, Wang Q. Enhanced recovery after surgery with laparoscopic radical gastrectomy for stomach carcinomas. World J Gastroenterol. 2015 Dec 21;21(47):13339-44. doi: 10.3748/wjg.v21.i47.13339. PMID 26715818
- [Background] Lee TG, Kang SB, Kim DW, Hong S, Heo SC, Park KJ. Comparison of early mobilization and diet rehabilitation program with conventional care after laparoscopic colon surgery: a prospective randomized controlled trial. Dis Colon Rectum. 2011 Jan;54(1):21-8. doi: 10.1007/DCR.0b013e3181fcdb3e. PMID 21160309
- [Background] van der Leeden M, Huijsmans R, Geleijn E, de Lange-de Klerk ES, Dekker J, Bonjer HJ, van der Peet DL. Early enforced mobilisation following surgery for gastrointestinal cancer: feasibility and outcomes. Physiotherapy. 2016 Mar;102(1):103-10. doi: 10.1016/j.physio.2015.03.3722. Epub 2015 May 7. PMID 26059985
- [Background] Havey R, Herriman E, O'Brien D. Guarding the gut: early mobility after abdominal surgery. Crit Care Nurs Q. 2013 Jan-Mar;36(1):63-72. doi: 10.1097/CNQ.0b013e3182753237. PMID 23221443